CLINICAL TRIAL: NCT05482035
Title: Clinical Trial on the Effectiveness of Blood Pressure Function of Wrist Blood Pressure Monitor
Brief Title: Clinical Trial of Wrist Blood Pressure Monitor in Conformance With the EN ISO 81060-2:2019/A1:2020 Standard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huawei Device Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-YBN2021075026A2
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure measured by wrist blood pressure monitor and mercury sphygmomanometer (Experimental)
  Interventions: Device: wrist blood pressure monitor

INTERVENTIONS:
Device: wrist blood pressure monitor — Comparing blood pressure measured by wrist blood pressure monitor with mercury sphygmomanometer .

SUMMARY:
The accuracy and safety of wrist blood pressure (model: MLY-B10) is evaluated according to the requirement of EN ISO 81060-2:2019/A1:2020.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should voluntarily participate in the clinical trial and sign the informed consent form.
2. Subjects must be willing and able to follow the investigation procedures.
3. Subjects are over 18 years old whose wrist circumference should be within 13.0-20.0 cm.

Exclusion Criteria:

1. Subjects with serious arrhythmias (atrial fibrillation, atrial flutter, ventricular flutter, ventricular fibrillation, ventricular tachycardia, borderline tachycardia, sinus arrest, pathological sinus syndrome, pacemaker rhythm) showed by electrocardiogram during screening period.
2. Subject with prior allergy to nylon, fluororubber, thermoplastic polyurethane elastomer (TPU), or polyvinyl chloride (PVC) materials.
3. Subjects with prior arterial obstructive disease or arteritis.
4. Subjects who had previously undergone mastectomy.
5. Subjects with wound or wrist inflammation were measured.
6. Subjects who are receiving intravenous infusion, blood transfusion, or other catheters at the site of measurement.
7. Subjects who had eaten, drank, smoked or exercised vigorously in the 30 minutes prior to the study.
8. Subjects who have participated in other clinical trials within 30 days that may affect this trial.
9. Subjects who the investigator consider inappropriate to attend the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
mean difference of systolic blood pressure | 30 minutes
  mean difference of systolic blood pressure between wrist blood pressure monitor and mercury sphygmomanometer
mean difference of diastolic blood pressure | 30 minutes
  mean difference of diastolic blood pressure between wrist blood pressure monitor and mercury sphygmomanometer
standard deviation of the difference of systolic blood pressure | 30 minutes
  standard deviation of the difference of systolic blood pressure between wrist blood pressure monitor and mercury sphygmomanometer
standard deviation of the difference of diastolic blood pressure | 30 minutes
  standard deviation of the difference of diastolic blood pressure between wrist blood pressure monitor and mercury sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen No.2 People's Hospital, Shenzhen, Guangdong, China